CLINICAL TRIAL: NCT05067283
Title: A Phase 1, Open-label, Multicenter Study to Assess Safety, Tolerability, PK, and Efficacy of MK-1084 as Monotherapy and as Part of Various Combination Therapies in Participants With KRAS G12C Mutant Advanced Solid Tumors
Brief Title: A Study of Calderasib (MK-1084) in KRAS Mutant Advanced Solid Tumors (MK-1084-001)
Acronym: KANDLELIT-001
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1084-001; MK-1084-001 (Other: MSD); jRCT2041220034 (Registry Identifier: jRCT); 2022-501563-40-00 (Registry Identifier: EU CT); U1111-1281-2482 (Registry Identifier: UTN)
Record Dates: First submitted 2021-10-01; First posted 2021-10-05 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — pembrolizumab; Carboplatin; Pemetrexed; Cetuximab; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Arm 1 (Experimental): Participants will receive daily oral escalating doses of up to 800 mg of calderasib until progressive disease or discontinuation. Dosing regimen may be adjusted based on safety.
  Interventions: Drug: Calderasib
- Arm 2 (Experimental): Participants will receive calderasib daily oral escalating dose of up to 800 mg plus pembrolizumab given as a 200 mg intravenous infusion once every 21-day cycle up to a total of 35 cycles (up to ~24 months). Treatment with calderasib will continue until progressive disease or discontinuation. Dosing regimen may be adjusted based on safety.
  Interventions: Drug: Calderasib; Biological: Pembrolizumab
- Arm 3 (Experimental): Participants will receive alternate formulation of calderasib until progressive disease or discontinuation. Dosing regimen may be adjusted based on safety.
  Interventions: Drug: Calderasib
- Arm 4 (Experimental): Participants will receive calderasib daily oral dose plus an intravenous infusion of pembrolizumab (200 mg) once every 21-day cycle for up to 35 cycles (up to ~24 months). Participants will also receive carboplatin (per label) and pemetrexed (per label) once every 21-day cycle for the first 4 cycles.
  Interventions: Drug: Calderasib; Biological: Pembrolizumab; Drug: carboplatin; Drug: pemetrexed
- Arm 5 (Experimental): Participants will receive calderasib daily oral dose plus an intravenous infusion of cetuximab (per label) every 2 weeks of each 28-day cycle.
  Interventions: Drug: Calderasib; Biological: cetuximab
- Arm 6 (Experimental): Participants will receive calderasib daily oral dose. Additionally, participants receive an intravenous infusion of cetuximab (per label) every 2 weeks of each 28-day cycle, oxaliplatin (per label) for first 6 cycles, and leucovorin (per label) and 5-fluorouracil (per label) once every 14-days.
  Interventions: Drug: Calderasib; Biological: cetuximab; Drug: oxaliplatin; Drug: leucovorin; Drug: 5-fluorouracil

INTERVENTIONS:
Drug: Calderasib — Oral dose
  Other Names: MK-1084
Biological: Pembrolizumab — Intravenous infusion of 200 mg
  Other Names: KEYTRUDA®; MK-3475
  Arms: Arm 2; Arm 4
Drug: carboplatin — Per label
  Arms: Arm 4
Drug: pemetrexed — Per label
  Arms: Arm 4
Biological: cetuximab — Per label
  Arms: Arm 5; Arm 6
Drug: oxaliplatin — Per label
  Arms: Arm 6
Drug: leucovorin — Per label
  Arms: Arm 6
Drug: 5-fluorouracil — Per label
  Arms: Arm 6

SUMMARY:
This is a study evaluating the safety, pharmacokinetics, and efficacy of calderasib alone, and calderasib plus other combination therapies in participants with advanced solid tumors with identified kirsten rat sarcoma viral oncogene homolog G12C (KRAS G12C) mutation.

ELIGIBILITY:
Inclusion Criteria:

For all participants:

* Has measurable disease by RECIST 1.1 criteria
* Has adequate organ function
* Male participants agree to protocol-specified contraception requirements including refraining from donating sperm and using protocol-specified contraceptives unless confirmed to be azoospermic
* Female participants must not be pregnant or breastfeeding, and must agree to protocol-specified contraceptive requirements and must have a negative highly sensitive pregnancy test within 24 hours (for a urine test) or 72 hours (for a serum test) before the first dose of study intervention

For Arm 1 - Has locally advanced unresectable or metastatic solid-tumor malignancy with histologically OR blood-based confirmation of KRAS G12C mutation who has received at least 1 line of therapy for systemic disease

For Arm 2

- Has an untreated metastatic non-small cell lung cancer (NSCLC) with histologically OR blood-based confirmation of KRAS G12C mutation and histologic confirmation of programmed cell death ligand 1 (PD-L1) tumor proportion score (TPS) ≥1%

For Arm 3

* Has locally advanced unresectable or metastatic solid-tumor malignancy with histologically or blood-based confirmation of KRAS G12C mutation who has received at least 1 line of therapy for systemic disease Expansion Group A: 2L+NSCLC
* Has histologically or cytologically confirmed diagnosis of unresectable or metastatic NSCLC with histological or blood-based confirmation of KRAS G12C mutation and submits archival tumor sample
* Previous treatment failure of at least 1 line of systemic therapy Expansion Group B
* Has locally advanced unresectable or metastatic solid-tumor malignancy, excluding NSCLC or CRC, with histologically or blood- based confirmation of KRAS G12C mutation who has received at least 1 line of therapy for systemic disease

Arm 4 only - Has an untreated advanced or metastatic nonsquamous NSCLC with histologically or blood-based confirmation of KRAS G12C mutation

Arm 5 only

* Histologically or cytologically confirmed diagnosis of locally advanced unresectable or metastatic colorectal adenocarcinoma and with histologically or blood-based confirmation of KRAS G12C mutation
* Previous treatment failure of one or 2 previous line(s) of systemic therapy

Arm 6 only

- Locally advanced unresectable or metastatic colorectal adenocarcinoma with histologically or blood-based confirmation of KRAS G12C mutation

Exclusion Criteria:

* Has received chemotherapy, definitive radiation, or biological cancer therapy within 4 weeks (2 weeks for palliative radiation) before first dose of study intervention
* Has a history of second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 5 years
* Has clinically active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has an active infection requiring systemic therapy
* Known history of HIV infection or. has a known history of Hepatitis B virus or known active Hepatitis C virus infection
* Has a history of interstitial lung disease, noninfectious pneumonitis requiring active steroid therapy, or ongoing pneumonitis
* Has an active autoimmune disease requiring systemic therapy
* Has not fully recovered from any effects of major surgical procedure without significant detectable infection
* Has one or more of the following ophthalmological findings/conditions: intraocular pressure >21 mm Hg and/or any diagnosis of glaucoma; diagnosis of central serous retinopathy, retinal vein occlusion, or retinal artery occlusion and/or a diagnosis of retinal degenerative disease
* Has received live or live-attenuated vaccine within 4 weeks of study start

Arm 4 Only

* Is unable to interrupt aspirin or other nonsteroidal anti-inflammatories (NSAIDs), other than an aspirin dose ≤1.3 grams per day, for at least 2 days (5 days for long-acting agents [for example, piroxicam]) before, during, and for at least 2 days after administration of pemetrexed.
* Is unable/unwilling to take folic acid, vitamin B12, and dexamethasone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 830 (Estimated)
Dates: Start 2021-12-17 (Actual); Primary Completion 2030-02-25 (Estimated); Study Completion 2030-02-25 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Experience a Dose-Limiting Toxicity (DLT) | Up to ~21 days
  A DLT is defined as an event with toxicity including the type, severity, time of onset, time of resolution, and the probable association with study treatment that are not due to pre-existing conditions as defined by the Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE 5.0). Number of participants who experience a DLT will be reported.
Number of Participants Who Experience an Adverse Event (AE) | Up to ~56 months
  An AE is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE. The number of participants who experience an AE will be reported.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to ~56 months
  An AE is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE. The number of participants who discontinue study treatment due to an AE will be reported.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to ~56 months
  ORR is defined as the percentage of participants who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1). The percentage of participants who experience a CR or PR as assessed by the investigator based on RECIST 1.1 will be reported.
Duration of Response (DOR) | Up to ~56 months
  DOR is defined as the time from first documented evidence of CR or PR until progressive disease (PD) or death. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. The DOR as assessed by the investigator will be reported.
Mean Plasma Concentration of calderasib | At designated timepoints during the study in Cycles 1, 2, 3, 5, 9, 13, 17, 21, 25, and every 6 weeks thereafter up to 56 months. Cycle=3 weeks (Arms 1-4) and 4 weeks (Arms 5-6)
  Mean Plasma Concentration of calderasib determined by blood samples collected pre-dose and at designated timepoints post-dose will be reported.
Maximum Concentration (Cmax) of calderasib | At designated timepoints during the study in Cycles 1, 2, 3, 5, 9, 13, 17, 21, 25, and every 6 weeks thereafter up to 56 months. Cycle=3 weeks (Arms 1-4) and 4 weeks (Arms 5-6).
  Cmax of calderasib determined by blood samples collected pre-dose and at designated timepoints post-dose will be reported.
Time to Maximum Concentration (Tmax) of calderasib | At designated timepoints during the study in Cycles 1, 2, 3, 5, 9, 13, 17, 21, 25, and every 6 weeks thereafter up to 56 months. Cycle=3 weeks (Arms 1-4) and 4 weeks (Arms 5-6)
  Tmax of calderasib determined by blood samples collected pre-dose and at designated timepoints post-dose will be reported.
Minimum Concentration (Cmin) of calderasib | At designated timepoints during the study in Cycles 1, 2, 3, 5, 9, 13, 17, 21, 25, and every 6 weeks thereafter up to 56 months. Cycle=3 weeks (Arms 1-4) and 4 weeks (Arms 5-6)
  Cmin of calderasib determined by blood samples collected pre-dose and at designated timepoints post-dose will be reported.
Area Under the Concentration Time-Curve 0-12 Hours (AUC 0-12) of calderasib | At designated timepoint during the study in Cycle 1 Day 1: Predose and up to 12 hours postdose. Cycle=3 weeks (Arms 1-4) and 4 weeks (Arms 5-6)
  AUC 0-12 of calderasib determined by blood samples collected pre-dose and at designated timepoints post-dose will be reported.
Area Under the Concentration Time-Curve 0-24 Hours (AUC 0-24) of calderasib | At designated timepoint during the study in Cycle 1 Day 1: Predose and up to 24 hours postdose. Cycle=3 weeks (Arms 1-4) and 4 weeks (Arms 5-6)
  AUC 0-24 of calderasib determined by blood samples collected pre-dose and at designated timepoints post-dose will be reported.
Half-Life (t1/2) of calderasib | At designated timepoint during the study in Cycle 1 Day 1: Predose and up to 24 hours postdose. Cycle=3 weeks (Arms 1-4) and 4 weeks (Arms 5-6)
  Half-Life (t1/2) of calderasib determined by blood samples collected pre-dose and at designated timepoints post-dose will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (73):
- United States (6):
  - Moffitt Cancer Center ( Site 0261), Tampa, Florida
  - START Midwest ( Site 0267), Grand Rapids, Michigan
  - John Theurer Cancer Center at Hackensack University Medical Center ( Site 0260), Hackensack, New Jersey
  - Laura and Isaac Perlmutter Cancer Center ( Site 0270), New York, New York
  - NEXT Virginia ( Site 0271), Fairfax, Virginia
  - MEDICAL COLLEGE OF WISCONSIN-Cancer Center Clinical Trials Office ( Site 0262), Milwaukee, Wisconsin
- Fundación CORI para la Investigación y Prevención del Cáncer ( Site 0438), La Rioja, Argentina
- Australia (4):
  - Chris O'Brien Lifehouse ( Site 0002), Camperdown, New South Wales
  - Liverpool Hospital-Medical Oncology ( Site 0001), Liverpool, New South Wales
  - Westmead Hospital ( Site 0006), Westmead, New South Wales
  - Monash Health-Oncology Research ( Site 0003), Clayton, Victoria
- Canada (5):
  - Cross Cancer Institute ( Site 0033), Edmonton, Alberta
  - The Moncton Hospital ( Site 0037), Moncton, New Brunswick
  - Hamilton Health Sciences-Juravinski Cancer Centre ( Site 0030), Hamilton, Ontario
  - Kingston Health Sciences Centre-Kingston General Hospital Site ( Site 0036), Kingston, Ontario
  - Princess Margaret Cancer Centre-Division of Medical Oncology and Hematology ( Site 0032), Toronto, Ontario
- Chile (4):
  - Centro de Estudios Clínicos SAGA-CECSAGA ( Site 0041), Santiago, Region M. de Santiago
  - FALP-UIDO ( Site 0040), Santiago, Region M. de Santiago
  - Bradfordhill ( Site 0042), Santiago, Region M. de Santiago
  - James Lind Centro de Investigacion del Cancer ( Site 0043), Temuco, Región de la Araucanía
- China (9):
  - Beijing Friendship Hospital Affiliate of Capital University-Oncology ( Site 0417), Beijing, Beijing Municipality
  - Fujian Cancer Hospital ( Site 0419), Fuzhou, Fujian
  - Southern Medical University Nanfang Hospital-Depatrment of Respiratory and Critical Care Medicine ( Site 0413), Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center-Internal medicine ( Site 0415), Guangzhou, Guangdong
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology ( Site 0418), Wuhan, Hubei
  - Jilin Cancer Hospital-oncology department ( Site 0412), Changchun, Jilin
  - Shanghai Chest Hospital-Oncology department ( Site 0410), Shanghai, Shanghai Municipality
  - Shanghai East Hospital ( Site 0416), Shanghai, Shanghai Municipality
  - Zhejiang Cancer Hospital-Thoracic oncology ( Site 0411), Hangzhou, Zhejiang
- Odense Universitetshospital-Department of oncology ( Site 0421), Odense, Region Syddanmark, Denmark
- Israel (5):
  - Rambam Health Care Campus-Oncology ( Site 0090), Haifa
  - Shaare Zedek Medical Center-Oncology ( Site 0092), Jerusalem
  - Hadassah Medical Center-Oncology ( Site 0094), Jerusalem
  - Meir Medical Center. ( Site 0091), Kfar Saba
  - Sheba Medical Center-ONCOLOGY ( Site 0093), Ramat Gan
- Italy (3):
  - Humanitas ( Site 0113), Rozzano, Lombardy
  - ospedale le scotte-U.O.C. Immunoterapia Oncologica ( Site 0111), Siena, Tuscany
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale ( Site 0110), Napoli
- Japan (5):
  - National Cancer Center Hospital East ( Site 0404), Kashiwa, Chiba
  - Kanagawa Cancer Center ( Site 0402), Yokohama, Kanagawa
  - Shizuoka Cancer Center ( Site 0401), Nakatogari, Shizuoka
  - National Cancer Center Hospital ( Site 0403), Chuo-ku, Tokyo
  - Cancer Institute Hospital of JFCR ( Site 0400), Koto, Tokyo
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kauno klinikos ( Site 0121), Kaunas, Kaunas County
  - Vilnius University Hospital Santaros Clinics Affiliate - National Cancer Center ( Site 0120), Vilnius
- Sarawak General Hospital ( Site 0453), Kuching, Sarawak, Malaysia
- New Zealand Clinical Research (Christchurch) ( Site 0004), Christchurch, Canterbury, New Zealand
- Panama (2):
  - Centro Oncologico de Panama ( Site 0160), Panama City
  - Centro Hemato Oncológico Paitilla ( Site 0163), Panama City
- Poland (4):
  - Uniwersytecki Szpital Kliniczny w Poznaniu ( Site 0172), Poznan, Greater Poland Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Oddzial Badan Wczesnych Faz ( Site 0170), Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne-Early Clinical Trials Unit ( Site 0171), Gdansk, Pomeranian Voivodeship
  - Oddzial Onkologii Klinicznej z Pododdzialem Chemioterapii Jednodniowej ( Site 0173), Koszalin, West Pomeranian Voivodeship
- South Korea (2):
  - Seoul National University Hospital ( Site 0191), Seoul
  - Samsung Medical Center-Division of Hematology/Oncology ( Site 0193), Seoul
- Spain (3):
  - Clinica Universidad de Navarra ( Site 0213), Madrid, Madrid, Comunidad de
  - Hospital Universitario Fundación Jiménez Díaz-START Madrid-FJD ( Site 0211), Madrid, Madrid, Comunidad de
  - Hospital Universitari Vall d'Hebron-Oncology ( Site 0212), Barcelona
- Switzerland (2):
  - Cantonal Hospital St.Gallen ( Site 0224), Sankt Gallen, Canton of St. Gallen
  - Ospedale Regionale Bellinzona e Valli ( Site 0220), Bellinzona, Canton Ticino
- Taiwan (3):
  - Chang Gung Memorial Hospital at Kaohsiung-Oncology and Hematology ( Site 0445), Kaohsiung Niao Sung Dist, Kaohsiung
  - National Cheng Kung University Hospital ( Site 0444), Tainan
  - National Taiwan University Hospital-Oncology ( Site 0443), Taipei
- Turkey (Türkiye) (4):
  - Ege University Medicine of Faculty ( Site 0231), Bornova, İzmir
  - Erciyes University ( Site 0232), Talas, Kayseri
  - Hacettepe Universite Hastaneleri-oncology hospital ( Site 0234), Ankara
  - Ankara City Hospital-oncology ( Site 0233), Ankara
- Ukraine (6):
  - MNPE ClinCenter of Oncology,Hematology,Transplantology and Palliative Care of CherkasyRegCouncil ( Site 0254), Cherkasy, Cherkasy Oblast
  - Communal Non-Commercial Enterprise Prykarpatski Clinical Onc-Chemotherapy department ( Site 0251), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Private Enterprise Private Manufacturing Company Acinus-Medical and Diagnostic Centre ( Site 0255), Kropyvnytskyi, Kirovohrad Oblast
  - Rivne Regional Clinical Hospital ( Site 0257), Rivne, Rivne Oblast
  - ME RIVNE REGIONAL ANTITUMOR CENTER ( Site 0259), Rivne, Rivne Oblast
  - Uzhhorod Multispecialty City Clinical Hospital ( Site 0258), Uzhhorod, Zakarpattia Oblast

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Derived] Ma X, Sloman DL, Duggal R, Anderson KD, Ballard JE, Bharathan I, Brynczka C, Gathiaka S, Henderson TJ, Lyons TW, Miller R, Munsell EV, Orth P, Otte RD, Palani A, Rankic DA, Robinson MR, Sather AC, Solban N, Song XS, Wen X, Xu Z, Yang Y, Yang R, Day PJ, Stoeck A, Bennett DJ, Han Y. Discovery of MK-1084: An Orally Bioavailable and Low-Dose KRASG12C Inhibitor. J Med Chem. 2024 Jul 11;67(13):11024-11052. doi: 10.1021/acs.jmedchem.4c00572. Epub 2024 Jun 26. PMID 38924388
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26313&tenant=MT_MSD_9011